CLINICAL TRIAL: NCT01342159
Title: Comparative Treatment of Intravitreal Bevacizumab and Triamcinolone Acetonide on Diabetic Macular Edema
Brief Title: Intravitreal Bevacizumab and Triamcinolone in Diabetic Macular Edema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hallym University Medical Center (Other)
Responsible Party: Hallym Medical Center, Hallym Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IVBITA; 20090321 (Other: Hallym Medical Center)
Record Dates: First submitted 2011-04-25; First posted 2011-04-27 (Estimated); Last update posted 2011-04-27 (Estimated); Status verified 2009-03

CONDITIONS: Diabetic Macular Edema
Keywords: bevacizumab, diabetic macular edema, triamcinolone
MeSH Terms: interventions — Intravitreal Injections

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Intravitreal bevacizumab injection (Active Comparator)
  Interventions: Procedure: Intravitreal injection
- Intravitreal Triamcinolone injection (Active Comparator)
  Interventions: Procedure: Intravitreal injection
- intravitreal bavacizumab with triamcinolone (Active Comparator)
  Interventions: Procedure: Intravitreal injection

INTERVENTIONS:
Procedure: Intravitreal injection — Intravitreal Injections were done under sterile conditions with topical anesthesia and insertion of a lid speculum. For the bevacizumab group, 1.25 mg (0.05 cc) bevacizumab (Avastin, made for F. Hoffmann-La Roche Ltd Basel, Switzerland by Genentech Inc., San Francisco, CA, USA) was injected intravitreally with a 30-gauge needle through the superotemporal quadrant. For the bevacizumab with triamcinolone group, in addition to intravitreal bevacizumab, 2 mg(0.05 cc) triamcinolone acetonide (Triamhexal, Hexal AG,Holzkirchen, Germany) was injected intravitreally through the inferotemporal quadrant. For triamcinolone group, 2 mg (0.05 cc) triamcinolone acetonide (Triamhexal, Hexal AG,Holzkirchen, Germany) was injected intravitreally.

SUMMARY:
One of the most frequent complications of diabetic retinopathy is diabetic macular edema. Recently, intravitreal bevacizumab and intravitreal triamcinolone were the most popular therapeutic modalities. However, as the long term effects of intravitreal bevacizumab and intravitreal triamcinolone on visual acuity and macular thickness have not been compared, it was the purpose of the present study to compare these treatment effects

DETAILED DESCRIPTION:
Randomization of intravitreal bevacizumab, intravitreal triamcinolone, intravitreal bevacizumab with triamcinolone on eyes with diabetic macular edema

ELIGIBILITY:
Inclusion Criteria:

* Diabetic macular edema (central macular thickness greater than 300 mm on optical coherence tomography )

Exclusion Criteria:

* history of glaucoma or ocular hypertension (defined as an intraocular pressure higher than 22 mmHg)
* an ocular condition (other than diabetes) that, in the opinion of the investigator, might affect macular oedema or alter visual acuity during the course of the study (e.g. retinal vein occlusion, uveitis or other ocular inflammatory disease, neovascular glaucoma, Irvine-Gass Syndrome, etc.)
* systemic corticosteroid therapy history of thromboembolic event (including myocardial infarction or cerebral vascular accident)
* major surgery within the prior 6 months or planned within the next 28 days

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-03; Primary Completion 2010-02 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Visual acuity | baseline, 1 month, 3 months, 6month, 9 month, 12 month

SECONDARY OUTCOMES:
Central macular thickness | baseline, 1 month, 3 months, 6 months, 12months
  analyzed by optical coherence tomography

CONTACTS AND LOCATIONS:
Locations (1):
- JiWon Lim, Chuncheon, South Korea